CLINICAL TRIAL: NCT01511952
Title: A Multi-Site Study of Music Therapy Interventions on Vitals, Feeding and Sleep in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: NICU Music Tx Interventions
Record Dates: First submitted 2012-01-16; First posted 2012-01-19 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Prematurity; Sepsis; SGA; RDS
Keywords: music therapy; entrainment; premature infants; live music intervention; parent preferred lullabies
MeSH Terms: conditions — Premature Birth; Sepsis | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Music intervention- SGA (Active Comparator): Infants will be randomly assigned to receive one of three music interventions randomized for the AM or PM
  Interventions: Other: Music Intervention; Other: Music
- Music Intervention- RDS (Active Comparator): Infants will be randomly assigned to receive music-one of 3 randomized interventions in the AM or PM
  Interventions: Other: Music Intervention; Other: Music
- Music Intervention- Sepsis (Active Comparator): Infants randomly assigned to receive one of three interventions-randomized for the AM or PM
  Interventions: Other: Music Intervention; Other: Music

INTERVENTIONS:
Other: Music Intervention — Applied by randomization-live at bassinet in the AM or PM Gato Box, Ocean Disc or parent-selected lullabies
Other: Music — Remo Ocean disc Gato box Music therapist's or Parent's preferred lullaby or 'Twinkle'
  Other Names: Remo Ocean disc; Gato box; Music therapist's or Parent's preferred lullaby or 'Twinkle'

SUMMARY:
This is a multi-site study of 272 premature infants >32 weeks who served in a randomized investigation (in morning or afternoon) where they served as their own controls. The infants' HR, RR, O2sats were measured with and without the implementation fo live music. The live interventions included songs of kin, selected by parents, the gato box and ocean disc played through entrained methods by a music therapist. The infants were evaluated within a two week period and in total each day including feeds, voids, activity level and sleep.

ELIGIBILITY:
Inclusion Criteria:

Premature infants diagnosed with SGA, RDS and/or Sepsis >32 weeks Referred by Neonatologist IRB HIPPA Informed Parent for infant consent obtained in writing

Exclusion Criteria:

Infants with diagnoses other than the above

Ages: 32 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 272 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The effects of live music intervention on premature baby function | over two weeks intervention periods
  Infants function according to flow sheet and in cumulative administration will be viewed with and without music therapy entrainment

SECONDARY OUTCOMES:
Vitals | 10 mins before, during and after intervention
  The HR, RR, O2sats, activity level, sleep. feeds and parental stress will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Joanne V Loewy, DA, MT-BC, LCAT, Principal Investigator — Beth Israel Medical Center